CLINICAL TRIAL: NCT00109616
Title: Newborn Antiseptic Washing and Neonatal Mortality-Nepal
Brief Title: Community Trial of Newborn Skin and Umbilical Cord Cleansing on Neonatal Mortality in Nepal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01HD044004 (NIH); R01HD044004 (NIH)
Record Dates: First submitted 2005-04-29; First posted 2005-05-02 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2006-01

CONDITIONS: Neonatal Mortality
Keywords: neonatal mortality; chlorhexidine; newborn cleansing; umbilical cord care; community-based trial; prevention trial; omphalitis
MeSH Terms: interventions — Soaps; Chlorhexidine

INTERVENTIONS:
Behavioral: Newborn skin cleansing with 0.25% chlorhexidine solution
Behavioral: Cleansing of umbilical cord with soap and water solution
Behavioral: Cleansing of umbilical cord with 4% chlorhexidine

SUMMARY:
Neonatal mortality and morbidity is common in Nepal and the vast majority of women deliver babies at home without a skilled birth attendant.

The purpose of this project is two-fold: 1) to evaluate whether washing a newborn child with a dilute antiseptic solution soon after birth can reduce mortality in the first 4 weeks of life and 2) to evaluate whether cleaning the umbilical cord and stump with either soap and water or an antiseptic solution for the first few days of life can reduce umbilical cord infections.

DETAILED DESCRIPTION:
While significant progress has been made in reducing preschool child mortality in developing countries over the past 20 years, much less progress has been made in reducing neonatal mortality and morbidity. Neonatal mortality rates are high in Nepal; a significant proportion of which are due to sepsis. In addition, the vast majority of women deliver babies at home without a skilled birth attendant and early neonatal care is routinely used in rural areas. Previous hospital-based research in Malawi suggested that newborn cleansing with a dilute chlorhexidine solution could reduce early infant mortality. This project evaluates the use of a simple intervention at the community level and the impact on neonatal mortality.

Comparisons: Two nested community-based randomized trials are being conducted. The first compares the neonatal mortality rates between newborn infants randomized to receive a whole body skin cleansing soon after birth with baby wipes impregnated with 0.25% chlorhexidine compared with newborns cleaned with baby wipes with a placebo solution. The second trial compares the rates of umbilical cord infections among children assigned to three groups:

* education of the mother on clean cord care alone;
* education of the mother plus routine washing of the cord and stump with soap and water solution for the first 10 days of life; -OR-
* education of the mother plus routine washing of the cord and stump with a 4% chlorhexidine solution.

Enrolled infants are visited on a regular basis during the first month of life to record vital status and grade the cord for signs of infection.

ELIGIBILITY:
Inclusion Criteria:

* All liveborn infants born in the study area

Exclusion Criteria:

* Newborn infants who died prior to study staff arriving to conduct the interventions

Ages: 1 Minute to 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 17000
Dates: Start 2002-10; Study Completion 2006-01

PRIMARY OUTCOMES:
neonatal mortality
umbilical cord infection

CONTACTS AND LOCATIONS:
Overall Officials: James M Tieslch, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States
- Nepal Nutrition Intervention Project-Sarlahi, Kathmandu and Sarlahi District, Nepal

REFERENCES:
- [Background] Mullany LC, Darmstadt GL, Tielsch JM. Role of antimicrobial applications to the umbilical cord in neonates to prevent bacterial colonization and infection: a review of the evidence. Pediatr Infect Dis J. 2003 Nov;22(11):996-1002. doi: 10.1097/01.inf.0000095429.97172.48. PMID 14614373
- [Background] Mullany LC, Darmstadt GL, Khatry SK, LeClerq SC, Tielsch JM. Safety of neonatal skin cleansing in rural Nepal. Indian Pediatr. 2006 Feb;43(2):117-24. PMID 16528107
- [Background] Mullany LC, Darmstadt GL, Tielsch JM. Safety and impact of chlorhexidine antisepsis interventions for improving neonatal health in developing countries. Pediatr Infect Dis J. 2006 Aug;25(8):665-75. doi: 10.1097/01.inf.0000223489.02791.70. PMID 16874163
- [Background] Mullany LC, Khatry SK, Sherchand JB, LeClerq SC, Darmstadt GL, Katz J, Gauchan P, Adhikari RK, Rana A, Tielsch JM. A randomized controlled trial of the impact of chlorhexidine skin cleansing on bacterial colonization of hospital-born infants in Nepal. Pediatr Infect Dis J. 2008 Jun;27(6):505-11. doi: 10.1097/INF.0b013e31816791a2. PMID 18449064
- [Result] Mullany LC, Darmstadt GL, Katz J, Khatry SK, Tielsch JM. Effect of instrument precision on estimation of low birth weight prevalence. J Perinatol. 2005 Jan;25(1):11-3. doi: 10.1038/sj.jp.7211209. PMID 15496868
- [Result] Mullany LC, Darmstadt GL, Khatry SK, Tielsch JM. Traditional massage of newborns in Nepal: implications for trials of improved practice. J Trop Pediatr. 2005 Apr;51(2):82-6. doi: 10.1093/tropej/fmh083. Epub 2005 Jan 26. PMID 15677372
- [Result] Mullany LC, Darmstadt GL, Khatry SK, Katz J, LeClerq SC, Shrestha S, Adhikari R, Tielsch JM. Topical applications of chlorhexidine to the umbilical cord for prevention of omphalitis and neonatal mortality in southern Nepal: a community-based, cluster-randomised trial. Lancet. 2006 Mar 18;367(9514):910-8. doi: 10.1016/S0140-6736(06)68381-5. PMID 16546539
- [Result] Mullany LC, Darmstadt GL, Katz J, Khatry SK, LeClerq SC, Adhikari RK, Tielsch JM. Development of clinical sign based algorithms for community based assessment of omphalitis. Arch Dis Child Fetal Neonatal Ed. 2006 Mar;91(2):F99-104. doi: 10.1136/adc.2005.080093. Epub 2005 Oct 13. PMID 16223755
- [Result] Mullany LC, Darmstadt GL, Coffey P, Khatry SK, LeClerq SC, Tielsch JM. A low cost, colour coded, hand held spring scale accurately categorises birth weight in low resource settings. Arch Dis Child. 2006 May;91(5):410-3. doi: 10.1136/adc.2005.088781. Epub 2006 Feb 7. PMID 16464960
- [Result] Mullany LC, Darmstadt GL, Khatry SK, LeClerq SC, Katz J, Tielsch JM. Impact of umbilical cord cleansing with 4.0% chlorhexidine on time to cord separation among newborns in southern Nepal: a cluster-randomized, community-based trial. Pediatrics. 2006 Nov;118(5):1864-71. doi: 10.1542/peds.2006-1091. PMID 17079556
- [Result] Mullany LC, Darmstadt GL, Katz J, Khatry SK, LeClerq SC, Adhikari RK, Tielsch JM. Risk factors for umbilical cord infection among newborns of southern Nepal. Am J Epidemiol. 2007 Jan 15;165(2):203-11. doi: 10.1093/aje/kwj356. Epub 2006 Oct 25. PMID 17065275
- [Result] Mullany LC, Darmstadt GL, Khatry SK, Leclerq SC, Tielsch JM. Relationship between the surrogate anthropometric measures, foot length and chest circumference and birth weight among newborns of Sarlahi, Nepal. Eur J Clin Nutr. 2007 Jan;61(1):40-6. doi: 10.1038/sj.ejcn.1602504. Epub 2006 Aug 2. PMID 16885929
- [Result] Tielsch JM, Darmstadt GL, Mullany LC, Khatry SK, Katz J, LeClerq SC, Shrestha S, Adhikari R. Impact of newborn skin-cleansing with chlorhexidine on neonatal mortality in southern Nepal: a community-based, cluster-randomized trial. Pediatrics. 2007 Feb;119(2):e330-40. doi: 10.1542/peds.2006-1192. Epub 2007 Jan 8. PMID 17210728
- [Result] Lee AC, Mullany LC, Tielsch JM, Katz J, Khatry SK, LeClerq SC, Adhikari RK, Shrestha SR, Darmstadt GL. Risk factors for neonatal mortality due to birth asphyxia in southern Nepal: a prospective, community-based cohort study. Pediatrics. 2008 May;121(5):e1381-90. doi: 10.1542/peds.2007-1966. PMID 18450881
- [Result] Rhee V, Mullany LC, Khatry SK, Katz J, LeClerq SC, Darmstadt GL, Tielsch JM. Maternal and birth attendant hand washing and neonatal mortality in southern Nepal. Arch Pediatr Adolesc Med. 2008 Jul;162(7):603-8. doi: 10.1001/archpedi.162.7.603. PMID 18606930
- [Result] Mullany LC, Katz J, Li YM, Khatry SK, LeClerq SC, Darmstadt GL, Tielsch JM. Breast-feeding patterns, time to initiation, and mortality risk among newborns in southern Nepal. J Nutr. 2008 Mar;138(3):599-603. doi: 10.1093/jn/138.3.599. PMID 18287373
- [Result] Lee AC, Mullany LC, Tielsch JM, Katz J, Khatry SK, LeClerq SC, Adhikari RK, Shrestha SR, Darmstadt GL. Verbal autopsy methods to ascertain birth asphyxia deaths in a community-based setting in southern Nepal. Pediatrics. 2008 May;121(5):e1372-80. doi: 10.1542/peds.2007-2644. PMID 18450880
- [Result] Sharma V, Katz J, Mullany LC, Khatry SK, LeClerq SC, Shrestha SR, Darmstadt GL, Tielsch JM. Young maternal age and the risk of neonatal mortality in rural Nepal. Arch Pediatr Adolesc Med. 2008 Sep;162(9):828-35. doi: 10.1001/archpedi.162.9.828. PMID 18762599
- [Result] Rosenberg RE, Ahmed S, Saha SK, Ahmed AS, Chowdhury MA, Law PA, Choi Y, Mullany LC, Tielsch JM, Katz J, Black RE, Santosham M, Darmstadt GL. Simplified age-weight mortality risk classification for very low birth weight infants in low-resource settings. J Pediatr. 2008 Oct;153(4):519-24. doi: 10.1016/j.jpeds.2008.04.051. Epub 2008 Jun 9. PMID 18539298
- [Result] Thatte N, Mullany LC, Khatry SK, Katz J, Tielsch JM, Darmstadt GL. Traditional birth attendants in rural Nepal: knowledge, attitudes and practices about maternal and newborn health. Glob Public Health. 2009;4(6):600-17. doi: 10.1080/17441690802472406. PMID 19431006
- [Result] Mullany LC, Darmstadt GL, Katz J, Khatry SK, Leclerq SC, Adhikari RK, Tielsch JM. Risk of mortality subsequent to umbilical cord infection among newborns of southern Nepal: cord infection and mortality. Pediatr Infect Dis J. 2009 Jan;28(1):17-20. doi: 10.1097/INF.0b013e318181fb4c. PMID 19034065
- [Result] Falle TY, Mullany LC, Thatte N, Khatry SK, LeClerq SC, Darmstadt GL, Katz J, Tielsch JM. Potential role of traditional birth attendants in neonatal healthcare in rural southern Nepal. J Health Popul Nutr. 2009 Feb;27(1):53-61. doi: 10.3329/jhpn.v27i1.3317. PMID 19248648
- [Result] Mullany LC, Katz J, Khatry SK, Leclerq SC, Darmstadt GL, Tielsch JM. Incidence and seasonality of hypothermia among newborns in southern Nepal. Arch Pediatr Adolesc Med. 2010 Jan;164(1):71-7. doi: 10.1001/archpediatrics.2009.239. PMID 20048245
- [Result] Karas DJ, Mullany LC, Katz J, Khatry SK, LeClerq SC, Darmstadt GL, Tielsch JM. Home care practices for newborns in rural southern Nepal during the first 2 weeks of life. J Trop Pediatr. 2012 Jun;58(3):200-7. doi: 10.1093/tropej/fmr057. Epub 2011 Jun 24. PMID 21705765
- [Result] Lee AC, Mullany LC, Tielsch JM, Katz J, Khatry SK, LeClerq SC, Adhikari RK, Darmstadt GL. Incidence of and risk factors for neonatal respiratory depression and encephalopathy in rural Sarlahi, Nepal. Pediatrics. 2011 Oct;128(4):e915-24. doi: 10.1542/peds.2010-3590. Epub 2011 Sep 26. PMID 21949140
- [Result] Lee AC, Mullany LC, Tielsch JM, Katz J, Khatry SK, Leclerq SC, Adhikari RK, Darmstadt GL. Community-based stillbirth rates and risk factors in rural Sarlahi, Nepal. Int J Gynaecol Obstet. 2011 Jun;113(3):199-204. doi: 10.1016/j.ijgo.2010.12.015. Epub 2011 Apr 1. PMID 21458812
- [Result] Mullany LC, Katz J, Khatry SK, LeClerq SC, Darmstadt GL, Tielsch JM. Neonatal hypothermia and associated risk factors among newborns of southern Nepal. BMC Med. 2010 Jul 8;8:43. doi: 10.1186/1741-7015-8-43. PMID 20615216
- [Result] Mullany LC, Katz J, Khatry SK, LeClerq SC, Darmstadt GL, Tielsch JM. Risk of mortality associated with neonatal hypothermia in southern Nepal. Arch Pediatr Adolesc Med. 2010 Jul;164(7):650-6. doi: 10.1001/archpediatrics.2010.103. PMID 20603466
- [Derived] Subedi S, Katz J, Erchick DJ, Verhulst A, Khatry SK, Mullany LC, Tielsch JM, LeClerq SC, Christian P, West KP, Guillot M. Does higher early neonatal mortality in boys reverse over the neonatal period? A pooled analysis from three trials of Nepal. BMJ Open. 2022 May 19;12(5):e056112. doi: 10.1136/bmjopen-2021-056112. PMID 35589346
- [Derived] Rosenstock S, Katz J, Mullany LC, Khatry SK, LeClerq SC, Darmstadt GL, Tielsch JM. Sex differences in neonatal mortality in Sarlahi, Nepal: the role of biology and environment. J Epidemiol Community Health. 2013 Dec 1;67(12):986-91. doi: 10.1136/jech-2013-202646. Epub 2013 Jul 19. PMID 23873992